CLINICAL TRIAL: NCT05050500
Title: Effects of Dapagliflozin on Inflammatory Factorslevel and Prognosis in Type 2 Diabetes With Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAFLO-CH; DAFLO (Registry Identifier: DAFLO-CH)
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction; Diabete Type 2; Glucose Intolerance
Keywords: myocardial infarction; dapagliflozin; MACE events
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — dapagliflozin; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Group (Experimental): Dapagliflozin 10 mg every 24 hours for 12 months
  Interventions: Drug: Dapagliflozin 10mg/Tab
- Control Group (Other): AMI standard therapy for 12 months
  Interventions: Drug: control group

INTERVENTIONS:
Drug: Dapagliflozin 10mg/Tab — patients meeting inclusion criteria will be randomized to receive dapagliflozin 10 mg every 24 hours for 6 months
  Other Names: Dapagliflozin Group
  Arms: Intervention Group
Drug: control group — patients meeting the inclusion criteria will be randomized to receive AMI standard therapy every 24 hours for 12 months.
  Arms: Control Group

SUMMARY:
Dapagliflozin is one of the SGLT-2 inhibiters. Recent clinical trials have demonstrated that SGLT-2 inhibitors are effective for treating heart failure. The DAPA-HF clinical trial has demonstrated that the effects of empagliflozin and dapagliflozin improve renal outcomes and reduce all-cause and cardiovascular death in patients with HFrEF[1]. However, its effect on myocardial infarction, the most common disease leading to death in the population, has not been evaluated sufficiently. A meta-analysis has demonstrated that compared with the control, SGLT2 inhibitor is associated with a reduction in the incidence of major adverse cardiovascular events (MACEs), myocardial infarction, cardiovascular mortality and all-cause mortality[2]. It seems that dapagliflozin might be effective for patients with acute myocardial infarction based on these studies. Thus, this study aims to evaluate the effect of dapagliflozin on short-term prognosis in patients with acute myocardial infarction compared to placebo.

1. Faiez Zannad, João Pedro Ferreira, Stuart J Pocock et el. SGLT2 inhibitors in patients with heart failure with reduced ejection fraction: a meta-analysis of the EMPEROR-Reduced and DAPA-HF trials. Lancet. 2020 Sep 19;396(10254):819-829.
2. Cai-Yan Zou, Xue-Kui Liu, Yi-Quan Sang et el. Effects of SGLT2 inhibitors on cardiovascular outcomes and mortality in type 2 diabetes: A meta-analysis. Medicine (Baltimore). 2019 Dec;98(49):e18245.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with acute MI, either STEMI or NSTEMI, according to the fourth universal definition of MI (Thygesen et al. 2019), disease onset within 7 days.
2. Previously diagnosed with type2 diabetes mellitus, newly diagnosed type2 diabetes according to ADA criteria or glucose intolerance.
3. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and the protocol.

Exclusion Criteria:

1. Patients diagnosed with Type 1 Diabetes Mellitus.
2. Patients with renal dysfunction. (GFR<90mmol/L).
3. Patients who have recently undergone immunosuppressive therapy.
4. Patients with a history of recurrent urinary tract infections.
5. Patients who are known to be allergic to SGLT-2 inhibitors.
6. Patients who are hemodynamically unstable.
7. Chronic symptomatic heart failure within the last year and known reduced ejection fraction (LVEF≤40 %), documented before the current MI hospitalization.
8. Severe hepatic impairment (Child-Pugh class C) at the time of inclusion into the trial.
9. Any other non cardiovascular diseases, such as active malignancy requiring treatment at the time of screening or with a life expectancy of fewer than two years based on the investigator´s clinical judgment.
10. Currently on treatment with a sodium-glucose co-transporter 2 inhibitor (SGLT2-inhibitor).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
MACE events | 12 months
  To assess the occurence of myocardial infarction, stroke and death from cardiovascular causes in post-infarction patients during the follow-up time.
Post-infarction angina | 12 months
  Evaluate the post-infarction angina occurence in both groups
The rate of heart failure occurrence | 12 months
  Assess the rate of new-onset heart failure during the study follow-up.
IL-6 | baseline, 1 month, 3 month, 6 month, 12 month
  Serum IL-6 level

SECONDARY OUTCOMES:
IL-1β | baseline, 1 month, 3 month, 6 month, 12 month
  Serum IL-1β
hs-CRP | baseline, 1 month, 3 month, 6 month, 12 month
  hs-CRP

CONTACTS AND LOCATIONS:
Overall Officials: Weisheng Liu, MD, Study Director — Qingdao Central Hospital
Locations (1):
- Mengmei Li, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No